CLINICAL TRIAL: NCT04334746
Title: The Discriminative Ability of the Four Balance Measures for.the Previous Fall Experience in Türkish Community-dwelling Older Adults
Brief Title: The Discriminative Ability of the Four Balance Measures for Fall History
Status: Completed | Type: Observational
Sponsor: Ordu University (Other)
Collaborators: Hacettepe University (Other); Giresun University (Other)
Responsible Party: Principal Investigator, Sevim ACARÖZ CANDAN, Department of Physiotherapy and Rehabilitation, Ordu University
Other Study IDs: OrduU8
Record Dates: First submitted 2020-04-02; First posted 2020-04-06 (Actual); Last update posted 2022-03-02 (Actual); Status verified 2022-03

CONDITIONS: Older People--Abuse of; Balance; Distorted; Fall

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Balance measurement tools — Timed Up and Go Test Functional Reach Test One-leg Stance Test Berg Balance Scale

SUMMARY:
The fall rate is increased parallel to the aging process. The early determination and management of falls in older adults are quite crucial to preserve the independence of older adults. In the literature, there are used many measurement tools for predicting fall status. The discriminative ability of these measures is important for the accuracy of the assessment. In this study, four of the most commonly used balance measurement tools will be investigated in terms of the discriminative ability for fall status in the Turkish community-dwelling older adults.

ELIGIBILITY:
Inclusion Criteria:

* being aged 65 or above,
* having a score of 21 or more from the Mini-Mental State Examination (MMSE) [20,23],
* able to ambulate independently or with an assistive device.

Exclusion Criteria:

* having visual and hearing problems that may cause restrictions in communication and also balance impairments,
* drug use (benzodiazepine, psychotropic drugs, etc.) with adverse effects on balance and walking,
* having any serious neurological, cardiopulmonary, or orthopedic disorders that adversely affected balance conditions.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Community-dwelling older adults
Sampling Method: Probability Sample
Enrollment: 351 (Actual)
Dates: Start 2020-10-06 (Actual); Primary Completion 2021-01-30 (Actual); Study Completion 2021-02-15 (Actual)

PRIMARY OUTCOMES:
Fall History | 2 minutes
  History of fallings will be determined through a question: "How many times have you fallen in the past year?".
  According to the participants' answers, the participants will be categorized into two groups: fallers (one or more fall events) and non-fallers (no falls).

SECONDARY OUTCOMES:
One-leg Stance test | 1 minute
  The static balance ability will be determined by one-leg stance test. The participants will be asked to stand on her/his dominant leg as long as possible. The standing time will be recorded with a stopwatch in seconds. Higher times indicate the better balance.
Berg Balance Scale | 20 minutes
  This scale will be used to evaluate the balance ability. It consists 14 items which are scored from 0 to 4, for a total score of 56 points possible. Higher scores indicate better balance performance.
Timed Up and Go Test | 3 minutes
  In this test, participants will be asked to stand from a chair, walk 3 meters (to a line on the floor), turn around, walk back to the chair, and sit back down. Participants are instructed to walk at a comfortable and safe pace during the Timed Up and Go Test. The participant's score is the time it takes to complete the mentioned test. Lower scores indicate better balance performance.
Functional Reach Test | 2 minutes
  Functional reach will be measured by using a leveled yardstick attached to the wall at the height of the participant's right acromion. To measure the participant's reaching distance, an examiner should stand 4 feet away from the yardstick and should be record the initial and end reach positions. Participant should stand in a relaxed position with feet approximately shoulder-width apart, made a loose fist, and, without touching the wall, placed the right arm parallel to the yardstick (initial position). Participants then will be asked to reach as far forward as they could without losing their balance (end position). The position of the third metacarpal along the yardstick will be recorded at both the initial and end positions. All subjects will be supervised during the test to ensure safety. The mean difference between the initial position and the end position will be calculated as the functional reach score in centimeters. The higher score indicates

CONTACTS AND LOCATIONS:
Overall Officials: Sevim Acaröz Candan, PhD, Study Director — Ordu University
Locations (1):
- Sevim ACARÖZ CANDAN, Ordu, Altinordu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No